CLINICAL TRIAL: NCT06292546
Title: The Effects of High-dose Dual Therapy Combined With Probiotics on Gut Microbiota for Helicobacter Pylori Rescue Treatment: A Prospective, Multicenter, Randomized Trial
Brief Title: The Effects of High-dose Dual Therapy With Probiotics on Gut Microbiota for Helicobacter Pylori Rescue Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Hospital (Xiamen), Fudan University (Other)
Responsible Party: Principal Investigator, Zhuyucheng, Deputy Chief Physician, Zhongshan Hospital (Xiamen), Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZYC-Hp2024
Record Dates: First submitted 2024-02-19; First posted 2024-03-05 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Gut Microbiota; Metabolic Disturbance; Helicobacter Pylori Eradication
Keywords: Helicobacter pylori; Eradication; Vonoprazan; Amoxicillin; Gut microbiota
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental): vonoprazan 20 mg bid + amoxicillin 0.75 g qid for 14 days, followed by 2 doses of bacillus subtilis enteric-coated capsules for 14 days.
  Interventions: Drug: Vonoprazan; Drug: Amoxicillin; Drug: Bacillus subtilis enteric-coated capsules
- Group B (Experimental): vonoprazan 20 mg bid + amoxicillin 0.75 g qid+ 2 doses of bacillus subtilis enteric-coated capsules for 14 days.
  Interventions: Drug: Vonoprazan; Drug: Amoxicillin; Drug: Bacillus subtilis enteric-coated capsules
- Group C (Experimental): 2 doses of bacillus subtilis enteric-coated capsules for 14 days, followed by vonoprazan 20 mg bid + amoxicillin 0.75 g qid for 14 days.
  Interventions: Drug: Vonoprazan; Drug: Amoxicillin; Drug: Bacillus subtilis enteric-coated capsules
- Group D (Active Comparator): vonoprazan 20 mg bid + amoxicillin 0.75 g qid for 14 days.
  Interventions: Drug: Vonoprazan; Drug: Amoxicillin

INTERVENTIONS:
Drug: Vonoprazan — Group A: vonoprazan 20 mg bid + amoxicillin 0.75 g qid for 14 days, followed by 2 doses of bacillus subtilis enteric-coated capsules for 14 days. Group B: vonoprazan 20 mg bid + amoxicillin 0.75 g qid+ 2 doses of bacillus subtilis enteric-coated capsules for 14 days. Group C: 2 doses of bacillus subtilis enteric-coated capsules for 14 days, followed by vonoprazan 20 mg bid + amoxicillin 0.75 g qid for 14 days. Group D: vonoprazan 20 mg bid + amoxicillin 0.75 g qid for 14 days.
Drug: Amoxicillin — Group A: vonoprazan 20 mg bid + amoxicillin 0.75 g qid for 14 days, followed by 2 doses of bacillus subtilis enteric-coated capsules for 14 days. Group B: vonoprazan 20 mg bid + amoxicillin 0.75 g qid+ 2 doses of bacillus subtilis enteric-coated capsules for 14 days. Group C: 2 doses of bacillus subtilis enteric-coated capsules for 14 days, followed by vonoprazan 20 mg bid + amoxicillin 0.75 g qid for 14 days. Group D: vonoprazan 20 mg bid + amoxicillin 0.75 g qid for 14 days.
Drug: Bacillus subtilis enteric-coated capsules — Group A: vonoprazan 20 mg bid + amoxicillin 0.75 g qid for 14 days, followed by 2 doses of bacillus subtilis enteric-coated capsules for 14 days. Group B: vonoprazan 20 mg bid + amoxicillin 0.75 g qid+ 2 doses of bacillus subtilis enteric-coated capsules for 14 days. Group C: 2 doses of bacillus subtilis enteric-coated capsules for 14 days, followed by vonoprazan 20 mg bid + amoxicillin 0.75 g qid for 14 days. Group D: vonoprazan 20 mg bid + amoxicillin 0.75 g qid for 14 days.
  Arms: Group A; Group B; Group C

SUMMARY:
The aim of this study was to evaluate the effects of High-dose Dual therapy combined with probiotics on the gut microbiota for Helicobacter pylori rescue treatment.

DETAILED DESCRIPTION:
The combination of vonoprazan (VPZ) and amoxicillin (VA therapy) has been shown to achieve notable eradication rates for Helicobacter pylori (H. pylori). Patients who receive this treatment are prone to adverse reactions, such as diarrhea, abdominal distention. We plan to combine probiotic with the above treatment. However, it is not clear what changes in gut microbiota and metabolism may result from this therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years;
* H.pylori infection diagnosed by 13C-urea breath test;
* A period of more than two months since the last eradication therapy for H. pylori;
* Patients who had previously failed 2 or more eradication regimens.

Exclusion Criteria:

* Allergy to any of the medications;
* Zollinger-Ellison syndrome, GC, Upper gastrointestinal bleeding, or Active peptic ulcer;
* Coexistence of significant concomitant illnesses, including heart disease, renal failure, hepatic disease, previous abdominal surgery, lactation, or pregnancy;
* Patients who had used probiotics, vonoprazan, and antibiotics in the past 12 weeks;
* Unwillingness to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Gut Microbiota | day 0, day 44 (or 58), day 104 (or 118)
  Diversity and Compositional Analysis of Gut Microbiota is tested by Metagenomics.

SECONDARY OUTCOMES:
Fecal Metabolites | day 0, day 44 (or 58), day 104 (or 118)
  Fecal metabolites is tested by Gas Chromatography-Mass Spectrometry Analysis.
Eradication rate | day 44 or day 58
  Eradication rate of H pylori, presenting with negative results on the 13C-UBT test.
Frequency of the adverse events | day 44 or day 58
  Incidence rate of the adverse events, including dyspepsia, nausea, vomiting, abdominal pain, bloating, diarrhea, dizziness, headache, skin rash, fatigue and fever.
Compliance rate of the drugs | day 44 or day 58
  Compliance is defined as good when they had taken more than 80% of the total medication.
Small intestinal bacterial overgrowth | day 0, day 44 (or 58), day 104 (or 118)
  Small intestinal bacterial overgrowth is tested by Hydrogen-Methane Breath.

CONTACTS AND LOCATIONS:
Overall Officials: Yucheng Zhu, Ph.D., Principal Investigator — Zhongshan Hospital (Xiamen), Fudan University
Locations (1):
- Zhongshan Hospital (Xiamen), Fudan University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No
We may balance the potential benefits and risks for each request and then provide the data that could be shared.

REFERENCES:
- [Result] Hu Y, Xu X, Ouyang YB, He C, Li NS, Xie C, Peng C, Zhu ZH, Shu X, Xie Y, Lu NH, Zhu Y. Altered Gut Microbiota and Short-Chain Fatty Acids After Vonoprazan-Amoxicillin Dual Therapy for Helicobacter pylori Eradication. Front Cell Infect Microbiol. 2022 Jun 2;12:881968. doi: 10.3389/fcimb.2022.881968. eCollection 2022. PMID 35719338